CLINICAL TRIAL: NCT02116959
Title: A Pilot Study Evaluating the Safety of Alternating Systemic Chemotherapy and Intra-Arterial Melphalan Chemotherapy in Children With Newly Diagnosed Advanced Intra-Ocular Retinoblastoma
Brief Title: Alternating Systemic Chemotherapy and Intra-Arterial Melphalan (IAM) Chemotherapy in Children With Intra-Ocular Retinoblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13087; NCI-2015-01749 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2014-02-18; First posted 2014-04-17 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Advanced Intra-Ocular Retinoblastoma; Retinoblastoma
Keywords: Systemic; Chemotherapy; Melphalan
MeSH Terms: conditions — Retinoblastoma | interventions — Melphalan; Carboplatin; Etoposide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients will receive alternating treatments beginning with systemic chemotherapy then followed by intra-arterial (IA) therapy.
  Bilateral retinoblastoma patients will be in Cohort 1.
  For bilateral Bilateral retinoblastoma patients where one eye is stage A or B and the other eye is C, D, or E, only the higher stage eye (C, D, E) will be treated with IA chemotherapy unless the stage A or B eye is not amenable or has failed local therapy.
  Interventions: Drug: Melphalan; Drug: Carboplatin; Drug: Etoposide; Drug: Vincristine
- Cohort 2 (Experimental): Patients will receive only intra-arterial (IA) therapy for more limited disease.
  Interventions: Drug: Melphalan; Drug: Carboplatin; Drug: Etoposide; Drug: Vincristine

INTERVENTIONS:
Drug: Melphalan
Drug: Carboplatin
Drug: Etoposide
Drug: Vincristine

SUMMARY:
The purpose of this study is to test the safety of the treatment combination of alternating standard chemotherapy and another (melphalan) chemotherapy at different interval schedules. Researchers want to find out what effects, good and/or bad, the treatment combination has on the patients and their retinoblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 3 months up to 18 years.
* Intraocular retinoblastoma not previously treated with systemic chemotherapy, radiation therapy, or IA therapy. Local retinal therapy such as laser photocoagulation and cryotherapy will be permitted.
* Unilateral or bilateral retinoblastoma (RB) patients are eligible
* Patients will be registered on study based on the local exam under anesthesia (EUA) done for diagnostic purposes prior to study entry. The EUA done at study entry should be done within 14 days prior to study entry
* Patients may have had enucleation of one eye, as long as the remaining eye meets the eligibility criteria
* Involved eye(s) must meet the definition for International Classification of Retinoblastoma
* For unilateral retinoblastoma (see Appendix 1 for International Classification of Retinoblastoma):

  1. Group A eye that has failed local therapy
  2. Group B eye that has failed local therapy
  3. Group C eye that has failed local therapy
  4. Group D eye
  5. Group E eye that is not buphthalmic, is not planned for enucleation after first cycle of chemotherapy, and is in a child less than 1 year of age
* For bilateral retinoblastoma (see Appendix 1 for International Classification of Retinoblastoma):

  1. Group A and Group A eyes that have failed local therapy
  2. Group A and Group B eyes that have failed local therapy
  3. Group A and Group C eyes
  4. Group A and Group D eyes
  5. Group A and Group E eyes in which the Group E eye is not planned for enucleation after first cycle of chemotherapy
  6. Group B and Group B eyes that have failed local therapy
  7. Group B and Group C eyes
  8. Group B and Group D eyes
  9. Group B and Group E eyes in which the Group E eye is not planned for enucleation after first cycle of chemotherapy
  10. Group C and Group C eyes
  11. Group C and Group D eyes
  12. Group C and Group E eyes even if early enucleation is planned for the Group E eye.
  13. Group D and Group D eyes
  14. Group D and Group E eyes even if early enucleation is planned for the Group E eye.
  15. Group E and Group E eyes if at least one eye is not planned for enucleation.
* Adequate Renal Function defined as: creatinine clearance or radioisotope Glomerular filtration rate (GFR) ³ 70 milliliter (mL)/min/1.73 m2 OR a serum creatinine based on age and gender derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the Center for Disease Control (CDC).
* Adequate hematological function defined as:

  1. Absolute Neutrophil Count > 1000/microliter
  2. Platelet Count > 100,000/microliter
* Adequate liver function defined as total bilirubin should be less than or equal to 1.5 x upper limit of normal (ULN) for age and serum glutamic-oxaloacetic transaminase (SGOT) / aspartate aminotransferase (AST) and serum glutamic-pyruvic transaminase (SGPT)

  / alanine aminotransferase (ALT) < 5 x upper limit of normal (ULN) for age
* Adequate coagulation system as defined as an international normalized ratio (INR) of less than 1.4 and a partial thromboplastin time (PTT) of less than 34
* Women and men of child-bearing potential must agree to use adequate contraception such as hormonal or barrier method of birth control or abstinence prior to study entry and for the duration of study participation. Should the subject or the subject's partner become pregnant or suspect pregnancy while on protocol therapy, the treating physician must be informed immediately.

Exclusion Criteria:

* Any evidence of extraocular retinoblastoma clinically or by magnetic resonance imaging (MRI) of brain and orbits with and without gadolinium. MRI may be done within 21 days prior to study entry.

  1. Evidence of systemic metastases on bilateral bone marrow, lumbar puncture, bone scan (or Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) scan), and/or any other additional tests done at study entry.
* Patients who have previously been treated with chemotherapy (with the exception of second inclusion criteria) radiation therapy, or intra-arterial therapy.
* Eyes with tumors that are amenable to local therapy with laser or cryotherapy without threat to vision
* Any technical factor that would prohibit use of catheterization of the ophthalmic artery (e.g., small for age infant, untreatable allergy to contrast).
* Abnormal cerebral vasculature noted on MR angiography that would increase the risk of the procedure, including but not limited to an incomplete Circle of Willis. Other abnormalities that are less severe than an incomplete Circle of Willis will be reviewed by the study chair in consultation with a neuro-interventional radiologist.
* Any serious ongoing condition, such as an untreated infection or organ dysfunction.
* Patients receiving any medications or substances that are inhibitors or inducers of CYP450 enzyme(s) are ineligible.
* Pregnant women are excluded from this study due to potential for teratogenic or abortifacient effects of therapy. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother breastfeeding should be discontinued upon start of protocol therapy.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Adverse Event evaluation for newly diagnosed advanced retinoblastoma treated with melphalan therapy and systemic chemotherapy | Up to 2 years
Dose-Limiting Toxicity (DLT) and minimum tolerated dosing interval for combination IAM and carboplatin, vincristine, and etoposide (CEV). | Up to 2 years

SECONDARY OUTCOMES:
Response rates after IAM combined with systemic CEV in patients with newly diagnosed advanced intraocular retinoblastoma | Up to 2 years
Ocular event free survival with the use of combination IAM therapy and systemic CEV in this patient population. | Up to 2 years
Visual outcomes using a standardized age based assessment | Up to 2 years
Salvage rate with triple IA therapy after failure of IA melphalan | Up to 2 years
Ocular event free survival for unilateral retinoblastoma with IA chemotherapy only for Group C or Group A/B that failed local therapy. | Up to 2 years
Visual outcomes using a standardized age based assessment. | Up to 2 years

OTHER OUTCOMES:
Collection of melphalan pharmacokinetics after intra-arterial administration to the retina | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Banerjee, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No